CLINICAL TRIAL: NCT00905476
Title: Analysis of the Prognosis and Clinical Course in Patients With Chronic Respiratory Failure Receiving Domiciliary NPPV
Brief Title: Prognosis in Patients With Chronic Respiratory Failure Receiving Domiciliary Noninvasive Positive Pressure Ventilation (NPPV)
Status: Completed | Type: Observational
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Toru Oga, Respiratory Care and Sleep Control Medicine, Kyoto University, Graduate School of Medicine, Kyoto University, Graduate School of Medicine
Other Study IDs: E552kyoto
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Respiratory Failure
Keywords: NPPV; Prognosis; Health-related quality of life; Patient reported outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NPPV: Patients with chronic respiratory failure receiving domiciliary NPPV

SUMMARY:
The purposes of the present study are (1) to analyze baseline patient characteristics cross-sectionally, (2) to analyze the prognosis and its predictive factors, and (3) to examine longitudinal clinical course in patients with chronic respiratory failure receiving domiciliary NPPV.

DETAILED DESCRIPTION:
Limited data are available about the prognosis and its predictive factors in patients with chronic respiratory failure receiving domiciliary NPPV. In addition, their health status, psychological status and sleep quality seem to be highly disturbed due to severe respiratory insufficiency. Therefore, in the present study, we aim to examine (1) contributive factors to health status based on baseline data, (2) whether patient reported measurements such as health status, dyspnea and psychological status would predict patient's future outcomes, and (3) how they would change for 3 years as compared to physiological measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic respiratory failure receiving domiciliary NPPV for more than 3 months

Exclusion Criteria:

* Uncontrolled severe comorbidities
* Patients with tracheotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic of respiratory medicine
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2009-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Prognosis/Mortality | 3 years

SECONDARY OUTCOMES:
Health status | At entry and every year for 3 years
Dyspnea | At entry and every year for 3 years
Psychological status | At entry and every year for 3 years
Sleep quality | At entry and every year for 3 years
Pulmonary function | At entry and every year for 3 years
Arterial blood gas | At entry and every year for 3 years
6 minute walking tests | At entry and every year for 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Chin, M.D., Study Chair — Graduate School of Medicine, Kyoto University
Locations (11):
- Japan (11):
  - NHO Minami-Kyoto Hospital, Jōyō
  - Kobe City Hospital Organization Medical Center West Hospital, Kobe
  - Kobe City Medical Center General Hospital, Kobe
  - Komaki Municipal Hospital, Komaki
  - Graduate School of Medicine, Kyoto University, Kyoto
  - Ogaki Municipal Hospital, Ōgaki
  - Otsu Red Cross Hospital, Ōtsu
  - Tosei General Hospital, Seto
  - Takatsuki Red Cross Hospital, Takatsuki
  - Tenri Hospital, Tenri
  - NHO Toneyama National Hospital, Toyonaka

REFERENCES:
- [Derived] Oga T, Taniguchi H, Kita H, Tsuboi T, Tomii K, Ando M, Kojima E, Tomioka H, Taguchi Y, Kaji Y, Maekura R, Hiraga T, Sakai N, Kimura T, Mishima M, Windisch W, Chin K. Comparison of Different Disease-Specific Health-Related Quality of Life Measurements in Patients with Long-Term Noninvasive Ventilation. Can Respir J. 2017;2017:8295079. doi: 10.1155/2017/8295079. Epub 2017 May 15. PMID 28588383